CLINICAL TRIAL: NCT00518232
Title: The Effective and Tolerable Titration Scheme and Dosage in Children With Attention-deficit Hyperactivity Disorder Treated With OROS-Methylphenidate
Brief Title: A Study to Determine Effective and Tolerable Titration Scheme for OROS-Methylphenidate in Children With Attention-deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Medical Director, Johnson & Johnson Taiwan, Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012508
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Methylphenidate; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: OROS-methylphenidate

SUMMARY:
The purpose of the study is to investigate the clinical benefit of switching children with ADHD from immediate-release methylphenidate (IR-MPH) to OROS-methylphenidate under the correct dosage conversion scheme.

DETAILED DESCRIPTION:
This is a prospective, non-comparative study. Each patient will be treated for 10 weeks including 6-week titration phase and 4-week maintenance phase. After an initial baseline evaluation, patients currently receiving IR-Methylphenidate (IR-MPH) therapy will switch to receiving OROS-methylphenidate once daily. Patients receiving IR-MPH =15 mg per day will switch to receive 18 mg once daily OROS-methylphenidate. For patients on IR-MPH daily dosage >15 mg and =30 mg, the initial dose of OROS-methylphenidate will be 36 mg once daily. Other patients receiving IR-MPH higher than 30 mg per day, will switch to receive 54 mg once daily OROS-methylphenidate. During the 6-week titration phase, those patients who do not achieve the criteria of "Optimal Response" will be titrated by biweekly increase to next dose level (36 mg per day, and then 54 mg per day). The maximum dose of OROS-methylphenidate per day is 54 mg as package insert indicates. However, dose decreases are allowed if clinically intolerable adverse events emerge. At the end of 6-week titration phase, the final titration dose should be maintained for the last 4 weeks of the trial regardless of the optimal response. In summary, all patients will attend bi-weekly clinic visits for the first 6 weeks (visit 2 to 4) and monthly clinic visits for the subsequent 4 weeks (visit 5). Patients will receive 18 mg or 36mg or 54 mg once daily OROS-methylphenidate for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who used to be treated their Attention-deficit hyperactivity disorder with IR-MPH less than 70 mg/day (inclusive) for at least one month without severe adverse events or possible contraindications with MPH
* Patients must be living with the parent/caregiver who can complete the questionnaires during the study
* Patients or parent/caregiver without any psychotic disease or any mental situation which may cause the concern to properly complete the questionnaires

Exclusion Criteria:

* Known to be non-responders to methylphenidate
* Marked anxiety, tension, aggression/agitation
* Known or suspected mental retardation or significant learning disorder
* Glaucoma, ongoing seizure disorder, psychotic disorder, diagnosis or family history of Tourette's disorder, bipolar disorder, eating disorder
* Subject who require drug therapy or hospitalization for treatment of a mood or anxiety disorder
* other psychotropic medication subject is taking at study entry could be continued during study period they were maintained at a stable dose for a minimum of 4 weeks pre-study entry

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 520 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To investigate the final dosage of OROS-methylphenidate for patients achieving optimal response in 10 weeks.The optimal response is defined as a score of 0 or 1 on each of the first 18 ADHD items (referred to SNAP-IV (Swanson, Nolan and Pelham))

SECONDARY OUTCOMES:
To describe the measurement of symptom(s)/sign(s) quality of life improvement and to describe the efficacy and the global assessment of satisfaction by parents/caregivers and patients at every visit throughout the study in 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd